CLINICAL TRIAL: NCT04058340
Title: The Effects of Taste Receptors Regulation in Upper Airway Innate Immunity of CF Patients
Brief Title: Taste Receptors Regulation in CF Patients
Acronym: CFTaste
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Lodz (Other)
Responsible Party: Principal Investigator, Pawel Majak, Principal Investigator, Medical University of Lodz
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: RNN/154/16/KE
Record Dates: First submitted 2019-08-12; First posted 2019-08-15 (Actual); Last update posted 2019-08-19 (Actual); Status verified 2019-08

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- lactizole-placebo (Active Comparator): A group of patients who will receive 3ml lactizole solution (150ppm) in nebulization twice a day for 4 weeks , and then for the next 4 weeks they will receive 2 times a day 3ml 0.9% NaCl solution in nebulization
  Interventions: Dietary Supplement: lactizole nebulization; Other: Placebo
- placebo-lactizole (Active Comparator): A group of patients who will receive 2 times a day for 4 weeks (0.9% NaCl solution in nebulization) for 4 weeks and will receive 3ml of lactizole solution (150ppm) in nebulization 2 times a day for 4 weeks
  Interventions: Dietary Supplement: lactizole nebulization; Other: Placebo

INTERVENTIONS:
Dietary Supplement: lactizole nebulization — Lactizole is generally recognized as safe: GRAS Flavor and Extract Manufacturers Association ( numer: 3773 ) Lactizole solution for nebulization was calculated based on dose-response curves; 150ppm was chosen as minimal effective (decreased sweet taste perception) and safety ( lack of FEV1 changes after nebulization)
Other: Placebo — 0.9% NaCl solution in nebulization

SUMMARY:
The project is intended to be realised in two phases. In the first stage, a case control study will be performed. In the second phase, double-blind, placebo controlled cross-over study will be conducted. The first stage it to compare innate immunity activation and Pseudomonas aeruginosa (Pa) expression between Pa positive and negative patients. In the second phase the effects of inhaled lactizole- TAS3R inhibitor will be assessed.

DETAILED DESCRIPTION:
Three visits have been planned during the entire study. During the first visit, all patients included in the study will have the following procedures: questionnaire tests, lung function tests, taste perception tests (gustometry) and exfoliative cytology of the nasal mucosa.

Patients with confirmed Pseudomonas aeruginosa presence in the airways will be randomly assigned to the Lactizole-Placebo group and the Placebo-Lactizole group, with a recommendation to take laktizol (3 ml) for 3 weeks at the concentration determined during the preliminary examination, in the nebulization 2 times per day) or placebo (3ml 0.9% NaCl solution in nebulization 2 once a day). The first nebulization of the solution issued during the visit will take place during the visit; each patient will undergo a clinical and spirometric assessment after 20 minutes of observation from completed nebulization.

During the second visit (after 4 weeks from visit 1), the first visit procedures will be repeated for all patients. Patients in the Lactizole-Placebo group will be recommended to take a placebo for 4 weeks (3 ml of 0.9% NaCl solution in nebulization 2 once a day); on the other hand, patients from the Placebo-Lactizole group will be advised to take lactisol for 4 weeks (3 ml of the solution in the concentration determined during the preliminary examination, in the nebulization 2 once a day). The first nebulization of the solution issued during the visit will take place during the visit; each patient will undergo a clinical and spirometric assessment after 20 minutes of observation from completed nebulization.

During the third visit (after 4 weeks from visit 2), the first visit procedures will be repeated for all patients.

ELIGIBILITY:
Inclusion Criteria:

* ulmonary manifestations of cystic fibrosis

Exclusion Criteria:

* first positive result of inoculation from the airways, which according to the standard is associated with the need for antibiotic therapy
* contraindication to a biopsy of the nasal mucosa
* exacerbation requiring antibiotics
* diabetes, exposure to tobacco smoke
* other chronic diseases and clinical conditions which, according to the researcher, may influence the assessed parameters and the course of the study.

Temporary exclusion criteria

- acute respiratory infection within 2 weeks from 1, 2 and 3 visits of the study.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-07-30 (Actual); Primary Completion 2019-11-30 (Estimated); Study Completion 2019-12-30 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Pseudomonas aeruginosa abundance | Change from Baseline after 4 weeks of the intervention
  Decrease of abundance of P. aeruginosa in throat swabs after nebulized lactizole . intervention. PCR testing for the presence of Pseudomonas aeruginosa genetic material (FTD Bacterial pneumoniae-HAP, Fast-track diagnostics Ltd., Malta)

SECONDARY OUTCOMES:
Change from Baseline in cystic fibrosis symptoms | Change from Baseline after 4 weeks of the intervention
  Questionnaire (standardized questionnaire to assess the degree of control of cystic fibrosis symptoms). Polish version of the Cystic Fibrosis Quality of Life Questionnaire (CFQoL) will be used
Change from Baseline in Lung function test | Change from Baseline after 4 weeks of the intervention
  Lung function test: spirometry will be performed in accordance with ERS / ATS standards
Change from Baseline in Taste perception | Change from Baseline after 4 weeks of the intervention
  Taste perception testing (gustometry): quantitative evaluation using a standardized TSTs diagnostic tool (Taste Strips, Burghart, Wedel, Germany
Change from Baseline in Nasal ILC1, 2 and 3 cells | Change from Baseline after 4 weeks of the intervention
  Nasal mucosa samples (Rhino-probe, ASI, Arlington, Texas). The assessment of the nasal mucosa material will include: percentage of ILC1, 2 and 3 cells (immunophenotyping and measurement by flow cytometry)
Change from Baseline in Nasal cytokines expression | Change from Baseline after 4 weeks of the intervention
  Nasal mucosa samples (Rhino-probe, ASI, Arlington, Texas). The assessment of the nasal mucosa material will include: mRNA expression for: Muc5b, Muc5ac, Beta-defensine, T1R3, T2Rs, selected cytokines (qPCR technique using self-designed primers)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Internal Medicine, Asthma and Allergy, Barlicki University Hospital, Medical University of Lodz, Lodz, Poland, Lodz, Poland

IPD SHARING:
Plan to Share IPD: No